CLINICAL TRIAL: NCT06822517
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1b Study of the NLRP3 Inhibitor VENT-02 in Patients With Mild to Moderate Parkinson's Disease
Brief Title: A Phase 1b Study of the NLRP3 Inhibitor VENT-02 in Patients With Mild to Moderate Parkinson's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Ventus Therapeutics U.S., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VENT-02-102
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VENT-02 Dose 1 (Experimental)
  Interventions: Drug: VENT-02
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VENT-02 — Orally administered capsules
  Arms: VENT-02 Dose 1
Drug: Placebo — Orally administered capsules
  Arms: Placebo

SUMMARY:
This trial is a randomized, double-blind, placebo-controlled Phase 1b study evaluating the safety/tolerability, PK, and pharmacodynamics of VENT 02, administered orally at 1 dose level twice daily (BID) over 28 days in patients with mild to moderate Parkinson's disease.

The study includes a screening period, a 28-day double-blind treatment period, and a 7-day follow-up period after last dose.

Approximately 30 patients will be randomized into 1 of the 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 90 years of age, inclusive.
* Body weight and body mass index (BMI) within the range of 100 to 265 pounds (45 to 120 kg) and 18 to 34 kg/m2 (inclusive), respectively.
* A diagnosis of idiopathic PD according to United Kingdom (UK) Brain Bank or Movement Disorder Society (MDS) criteria with bradykinesia and ≥ 1 additional cardinal sign of PD (e.g., resting tremor, rigidity).
* A diagnosis of PD for ≤ 7 years at Screening.
* A modified Hoehn & Yahr stage 1 to 2.5.
* If presently receiving treatment for PD, must be on a stable dose for ≥ 2 weeks prior to dosing, with no expected change in this regimen for the duration of the study.
* If presently taking any non-PD concomitant medications, must be on a stable dose for ≥ 2 weeks prior to dosing.

Exclusion Criteria:

* Any clinically significant abnormality at Screening
* A positive serology for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV) 1/2 at Screening.
* A significant neurological disease affecting the central nervous system, other than PD, that may affect cognition or ability to complete the study, including but not limited to dementias, severe and repetitive past (up to 5 years) head trauma, normal pressure hydrocephalus, or epilepsy or recurrent seizures (except febrile childhood seizures), as determined by the investigator.
* Current serious or unstable illnesses, that, in the investigator's opinion, could compromise patient safety and ability to comply with study procedures, or has a life expectancy of < 24 months.
* A history of suicidal ideation or previous suicide attempt in the 12 months prior to Screening or is clinically judged by the investigator to be at serious risk for suicide as assessed by medical history, examination, or the C-SSRS.
* A contraindication (e.g., current use of anticoagulants) that would prohibit a lumbar puncture (LP).
* Currently enrolled in any other interventional clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study, as assessed by the investigator.
* Has participated in a clinical trial involving an investigational product within 30 days or 5 half-lives (whichever is longer) prior to dosing.
* Has levodopa-induced dyskinesias lasting for > 25% of waking day or dyskinesias interfering with many daily activities.
* Has dysphagia to the extent that it would affect the patient's ability to swallow the investigational medicinal product (IMP).
* Has a parkinsonian syndrome, including atypical parkinsonism.
* Is a known carrier (i.e., confirmed by historical medical documentation) of familial PD genes.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to Follow-up Visit (Day 35)
  Number of treatment-emergent adverse events (TEAEs) with VENT-02 treatment compared to placebo

SECONDARY OUTCOMES:
Concentrations of biomarkers | Baseline to Day 28
  Change from baseline in concentrations of biomarkers of inflammation and neurodegeneration in plasma and CSF
Concentrations of VENT-02 in plasma and CSF | Baseline to Day 28
  PK as measured by concentrations of VENT-02 in plasma and CSF

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Investigative Site, Fountain Valley, California
  - Investigative Site, San Jose, California
  - Investigative Site, West Hills, California
  - Investigative Site, Englewood, Colorado
  - Investigative Site, Aventura, Florida
  - Investigative Site, Boca Raton, Florida
  - Investigative Site, Coral Gables, Florida
  - Investigative Site, Coral Springs, Florida
  - Investigative Site, Cutler Bay, Florida
  - Investigative Site, Daytona Beach, Florida
  - Investigative Site, Doral, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Maitland, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Winter Park, Florida
  - Investigative Site, Scarborough, Maine
  - Investigative Site, Farmington Hills, Michigan
  - Investigative Site, Abington, Pennsylvania
  - Investigative Site, Memphis, Tennessee
  - Investigative Site, Cypress, Texas
  - Investigative Site, Round Rock, Texas
  - Investigative Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No